CLINICAL TRIAL: NCT04476992
Title: A Safety Study on the Use of Intermittent Versus Continuous Inhalation of NO in Spontaneous Breathing COVID-19 Patients
Brief Title: Nitric Oxide Therapy for COVID-19 Patients With Oxygen Requirement
Acronym: NICOR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Siberian State Medical University (Other)
Responsible Party: Principal Investigator, Nikolay Kamenshchikov, Medical Doctor, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICOR
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Hypoxemia; Pneumonia, Viral; Coronavirus Infection
Keywords: Nitric Oxide gas; COVID-19; Hypoxemia; Viral Pneumonia
MeSH Terms: conditions — Hypoxia; Pneumonia, Viral; Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NO High Concentration (Active Comparator): Nitric oxide will be delivered twice a day with a non-rebreathing system that allows a safe administration of Nitric Oxide gas at high concentrations limiting the amount of NO2 delivered to the patient.
  Interventions: Drug: Nitric Oxide-Sessions
- NO High Concentration + Continuous Low Concentration (Experimental): Nitric oxide will be delivered twice a day with a non-rebreathing system that allows a safe administration of Nitric Oxide gas at high concentrations limiting the amount of NO2 delivered to the patient.
  This arm will receive in addition a continuous low flow of Nitric Oxide at 20 ppm among the high concentration treatments.
  Interventions: Drug: Nitric Oxide-Continuous and Sessions

INTERVENTIONS:
Drug: Nitric Oxide-Sessions — Nitric Oxide will be delivered at 200 ppm in 2 daily sessions (morning, evening; 9-12 hours apart) for 14 days. Each session will last 30 minutes, for a total of 60 minutes/day for each patient. A tank of NO gas will be connected to the inspiratory limb of the circuit, and the flow will be adjusted to deliver a target concentration of 200 ppm NO. Commercially available tanks will be used to provide the gas. The desired mixture of air, oxygen (O2), and NO will be titrated with the respective flowmeter to reach a concentration of 200 ppm at the inspiratory limb with the desired Fraction of inspired oxygen (FiO2).
  Other Names: Nitric Oxide inhalation at high concentration
  Arms: NO High Concentration
Drug: Nitric Oxide-Continuous and Sessions — Nitric Oxide will be delivered at 200 ppm in 2 daily sessions (morning, evening; 9-12 hours apart) for 14 days. Each session will last 30 minutes, for a total of 60 minutes/day for each patient. A tank of NO gas will be connected to the inspiratory limb of the circuit, and the flow will be adjusted to deliver a target concentration of 200 ppm NO. Commercially available tanks will be used to provide the gas. The desired mixture of air, oxygen (O2), and NO will be titrated with the respective flowmeter to reach a concentration of 200 ppm at the inspiratory limb with the desired Fraction of inspired oxygen (FiO2).
  The subjects assigned to the group "NO High Concentration + Continuous Low Concentration" will receive in adjunction a continuous dose of NO at 20 ppm.
  Other Names: Nitric Oxide inhalation at high concentration + low concentration
  Arms: NO High Concentration + Continuous Low Concentration

SUMMARY:
Preliminary data support the effect of Nitric Oxide (NO) on improving the oxygenation in mechanically ventilated patients and spontaneously breathing patients with COVID-19. In vitro studies showed an antiviral effect of NO against SARS-coronavirus. The optimal therapeutic regimen of NO gas in spontaneously breathing hypoxemic patients with COVID-19 is not known. We hypothesize that high concentration inhaled NO with an adjunct of continuous low dose administration between the high concentration treatments can be safely administered in hypoxemic COVID-19 patients compared to the high dose treatment alone. Prolonged administration of NO gas may benefit the patients in terms of the severity of the clinical course and time to recovery. Together with a clinical effect on ventilation-perfusion matching, a prolonged regimen would allow also an increase in antiviral activity (dose and time-dependent).

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) consists mainly of a respiratory infection that spans from a mild involvement of the upper respiratory tract to severe pneumonia leading to respiratory distress, shock, and death. Fever, cough, and dyspnea/tachypnea, together with myalgia and fatigue, have been identified as the most common presenting symptoms. Most of the patients remain in a state of mild upper respiratory tract disease for a relatively long period (a median of 8-10 days), after which a proportion of up to 25% may develop severe hypoxemia and ARDS with the necessity of mechanical ventilation. Deterioration with ICU admission (most likely in older patients with comorbidities) raises the incidence of mortality in a range that goes from 3.4 up to 61%. Moreover, ICU admission poses a significant strain in terms of healthcare resources. Thus, a treatment able to avoid the progression of the disease from the mild to the severe phases would have a substantial benefit both in terms of lives saved and hospital resources spared. However, at the time, only Remdesivir and Dexamethasone have shown some benefits in robust clinical trials.

Nitric Oxide gas is a therapy currently approved for the treatment of pulmonary hypertension in newborns and is also used as rescue therapy in patients with acute respiratory distress syndrome (ARDS). The clinical role of NO gas in COVID-19 patients could be of particular relevance since there is in-vitro evidence of NO antiviral activity specifically against SARS coronavirus. At the time of the SARS pandemic, a small rescue trial on intubated patients with SARS showed that NO was effective in improving the oxygenation, fasten the resolution of chest X-ray abnormalities, and improve the clinical outcomes. Moreover, in vitro studies demonstrated that the NO-donor compound S-nitroso-N-acetylpenicillamine was able to increase the survival rate of in vitro mammalian cells infected with SARS-CoV. SARS-CoV and SARS-CoV-2 share the same subgenus inside the family Coronaviridae. The literature seems to point towards an a-specific rather than pathogen-specific antimicrobial effect of NO. Thus, the role of exogenous inhaled NO as a viricidal agent during COVID-19 infection could be hypothesized.

Nitric Oxide at high concentration has been found to be microbicidal but still safe in spontaneously breathing subjects in a phase I trial. There are several trials testing the efficacy of NO therapy in improving the outcome of COVID-19 patients. So far, only a retrospective observational study showed that NO gas is useful in improving the oxygenation in spontaneously breathing patients. However, the optimal therapeutic regimens and the efficacy of NO gas in improving the oxygenation in hypoxemic COVID-19 patients haven't been tested.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 confirmed by a positive RT-PCR test
* Hospital admission within 11 days from the onset of symptoms
* Spontaneous breathing with oxygen requirement ≥1 L/min
* Expected discharge > 96 hours at randomization

Exclusion Criteria:

* Pregnancy
* Presence of a tracheostomy
* Assistance by any non-invasive CPAP or NIV at the screening
* Treatment with high flow nasal cannula at the screening
* Clinical contraindication to the use of NO
* Patients enrolled in another interventional trial
* Hospitalized and confirmed diagnosis of COVID-19 for more than 7 days
* Previous intubation for COVID-19
* Subject not committed to full support (DNR, DNI or CMO)
* Subject requiring oxygen at home for lung comorbidities
* The primary cause of hospitalization not due to COVID-19
* Subject receiving vasopressor at the time of screening
* History of malignancy or other irreversible disease/conditions with 6-month mortality >50%
* Oxygen saturation of 100% at screening, despite oxygen requirement
* Patients on dialysis at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Methemoglobin level at 48 hours | 48 hours
  The primary outcome will be evaluated with the difference in Methemoglobin levels between the groups at 48 hours after randomization.

SECONDARY OUTCOMES:
Change in Methemoglobin level at 96 hours | 96 hours
  The primary outcome will be evaluated with the difference in Methemoglobineamia between the groups at 96 hours after randomization.
Improvement in oxygenation between the groups at 48 hours or at discharge if before 48 hours | 48 hours
  The secondary outcome, "Improve the oxygenation at 48 hours," will be evaluated with the measure of the difference in oxygenation among the groups at 48 hours. Oxygenation will be measured in terms of the SpO2/FiO2 ratio.
Improvement in oxygenation between the groups at 96 hours or at discharge if before 96 hours | 96 hours
  The secondary outcome, "Improve the oxygenation at 96 hours," will be evaluated with the measure of the difference in oxygenation between the groups at 96 hours. Oxygenation will be measured in terms of the SpO2/FiO2 ratio.
Rate of positive RT-PCR for SARS-CoV-2 between groups in 5 days, discharge, and 28 days | 28 days
  The secondary outcome "difference in the rate of negative RT-PCR for SARS CoV-2" will be evaluated as the rate of negativization of the RT-PCR for SARS-CoV-2 at 5 days after randomization, at discharge and at 28 days after randomization.
Time to clinical recovery among groups, defined as time to interruption of oxygen administration for 24 hours or discharge | 28 days
  The secondary outcome "different time to clinical recovery" will be evaluated as the time between the randomization and the clinical indication to interrupt the administration of oxygen for 24 hours.
Reduction in the inflammatory markers among groups | 7 days
  The secondary outcome "Different reduction in inflammatory markers" will be evaluated as improvement in the inflammatory markers (IL-6; Ferritin; White Blood Cells; Leucocyte count; CRP; D-Dimer) observed in blood samples collected at day 1, 2, 3, 4, and 7 compared to the Baseline value.
Rate of Acute Kidney Disease (AKI) between groups during hospitalization | 28 days
  The secondary outcome "rate of AKI between groups" will be evaluated as the presence of a comparable rate of AKI during the hospital stay. The AKI will be defined according to the KDIGO classification.
Difference in Katz score between groups | 28 days
  The secondary outcome "Difference in Katz score between groups" will be evaluated as the difference in Katz Activities of Daily Living between Baseline and day 28. This questionnaire will coincide with the 28-day phone call to assess health status and survival.

OTHER OUTCOMES:
Effect of NO gas treatment on cardiovascular hemodynamics assessed using cardiac ultrasound in COVID-19 hypoxemic patients | 96 hours
  1. The exploratory outcome "Effect of nitric oxide on heart function in COVID-19 hypoxemic patients" will be evaluated as:
  1. the changes observed in heart ultrasound at 48 and 96 hours (or at discharge) compared to the Baseline in all groups.
  2. the changes observed in heart ultrasound during the administration of NO comparing pre-treatment, during treatment, and post-treatment.
Effect of NO gas treatment on lung function evaluated with serial spirometry in COVID-19 hypoxemic patients | 96 hours
  2. The secondary outcome "Effect of NO gas on lung function in COVID-19 hypoxemic patients" will be evaluated as:
  1. the changes observed in spirometry at 48 and 96 hours (or at discharge) compared to the Baseline in all groups.
  2. the changes observed in spirometry during the administration of NO comparing pre-treatment, during treatment, and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay O Kamenshchikov, M.D., Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia

REFERENCES:
- [Derived] Kamenshchikov NO, Safaee Fakhr B, Kravchenko IV, Dish AY, Podoksenov YK, Kozlov BN, Kalashnikova TP, Tyo MA, Anfinogenova ND, Boshchenko AA, Berra L. Assessment of continuous low-dose and high-dose burst of inhaled nitric oxide in spontaneously breathing COVID-19 patients: A randomized controlled trial. Nitric Oxide. 2024 Aug 1;149:41-48. doi: 10.1016/j.niox.2024.06.003. Epub 2024 Jun 14. PMID 38880198